CLINICAL TRIAL: NCT02716116
Title: A Phase 1/2 Study of the Safety, Pharmacokinetics, and Anti-Tumor Activity of the Oral EGFR/HER2 Inhibitor TAK-788 (AP32788) in Non-Small Cell Lung Cancer
Brief Title: A Study of TAK-788 in Adults With Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP32788-15-101; U1111-1217-7205 (Registry Identifier: WHO); 2016-001271-68 (EudraCT Number)
Record Dates: First submitted 2016-03-14; First posted 2016-03-23 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — mobocertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1: Dose Escalation Component (Experimental): TAK-788 treatment for participants with advanced NSCLC.
  Interventions: Drug: TAK-788
- Part 2: Expansion Cohort 1 (Experimental): TAK-788 treatment for NSCLC participants with EGFR exon 20 activating insertions, who have either not received or not shown an objective response to an EGFR tyrosine kinase inhibitors (TKI), and who have no active, measurable central nervous system (CNS) metastases.
  Interventions: Drug: TAK-788
- Part 2: Expansion Cohort 2 (Experimental): TAK-788 treatment for NSCLC participants with HER2 exon 20 activating insertions or point mutations and no active, measurable CNS metastases.
  Interventions: Drug: TAK-788
- Part 2: Expansion Cohort 3 (Experimental): TAK-788 treatment for NSCLC participants with EGFR exon 20 activating insertions or HER2 exon 20 activating insertions or point mutations and active, measurable CNS metastases.
  Interventions: Drug: TAK-788
- Part 2: Expansion Cohort 4 (Experimental): TAK-788 treatment for NSCLC participants with other targets against which TAK-788 is active (examples include EGFR exon 19 deletions or exon 21 substitutions [with or without T790M mutations] and other uncommon EGFR activating mutations), without active CNS metastases.
  Interventions: Drug: TAK-788
- Part 2: Expansion Cohort 5 (Experimental): TAK-788 treatment for NSCLC participants with EGFR exon 20 activating insertions, who have previously shown an objective response to an EGFR TKI and subsequently progressed without active CNS metastases.
  Interventions: Drug: TAK-788
- Part 2: Expansion Cohort 6 (Experimental): TAK-788 treatment NSCLC participants with EGFR exon 20 activating insertions, who have not received prior systemic anticancer treatment for locally advanced or metastatic disease without active CNS metastases
  Interventions: Drug: TAK-788
- Part 2: Expansion Cohort 7 (Experimental): TAK-788 treatment for participants with solid tumors other than NSCLC with EGFR/HER2 mutations against which TAK-788 is active without active CNS metastases.
  Interventions: Drug: TAK-788
- Part 3: Extension Cohort (Experimental): TAK-788 treatment for participants with previously treated locally advanced or metastatic NSCLC whose tumors harbor EGFR exon 20 insertion mutations.
  Interventions: Drug: TAK-788

INTERVENTIONS:
Drug: TAK-788 — TAK-788 capsules.
  Other Names: AP32788

SUMMARY:
This study is about a medicine called TAK-788, also known as mobocertinib, given to adults with non-small cell lung cancer. The main aims of this study are to check if there are any side effects from TAK-788, to learn how TAK-788 is processed by the body, and to determine the best dose of TAK-788 to treat this condition. Participants will take TAK-788 capsules with chemotherapy. Participants will continue to take TAK-788 unless they or their doctor decide they should stop this treatment. Participants will take TAK-788 capsules with or without chemotherapy under antidiarrhea prevention to determine the safety of TAK-788 treatment. Non-Asian, non-White participants will take TAK-788 to determine the safety and tolerability of TAK-788 treatment.

DETAILED DESCRIPTION:
This phase 1/2 study will evaluate the safety, pharmacokinetics, and anti-tumor activity of oral EGFR/HER2 Inhibitor TAK-788 in participants with NSCLC and anti-tumor activity of TAK-788 in participants with solid tumors other than NSCLC with EGFR or HER2 mutations. The trial will be conducted in three parts: a dose escalation (Part 1), expansion phase (Part 2), followed by an extension phase (Part 3).

The objectives of the dose escalation phase (Part 1), is to determine the safety profile of orally administered TAK-788, including the MTD, DLTs, RP2D, pharmacokinetic profile. The primary goal of the expansion component of the trial is to evaluate the anti-tumor activity of TAK-788 in seven histologically and molecularly defined cohorts at the RP2D (determined based on dose escalation phase of the trial).

The seven expansion cohorts will be:

1. NSCLC participants with EGFR exon 20 activating insertions, who have either not received or not shown an objective response to an EGFR TKI, and who have no active, measurable CNS metastases;
2. NSCLC participants with HER2 exon 20 activating insertions or point mutations and no active, measurable CNS metastases;
3. NSCLC participants with EGFR exon 20 activating insertions or HER2 exon 20 activating insertions or point mutations and active, measurable CNS metastases;
4. NSCLC participants with other targets against which TAK-788 is active (examples include EGFR exon 19 deletions or exon 21 substitutions [with or without T790M mutations] and other uncommon EGFR activating mutations), without active CNS metastases;
5. NSCLC participants with EGFR exon 20 activating insertions, who have previously shown an objective response to an EGFR TKI and subsequently progressed, without active CNS metastases;
6. NSCLC participants with EGFR exon 20 activating insertions, who have not received prior systemic anticancer treatment for locally advanced or metastatic disease, without active CNS metastases; and
7. Participants with solid tumors other than NSCLC with EGFR/HER2 mutations against which TAK-788 is active, without active CNS metastases.

The extension phase will evaluate efficacy of TAK-788 in participants with locally advanced or metastatic NSCLC whose tumors harbor EGFR exon 20 insertion mutations and who have been previously treated. The study enrolled 324 participants.

ELIGIBILITY:
General Inclusion Criteria all cohorts: dose escalation, antidiarrhea prophylaxis, dose escalation combination, expansion, and extension:

1. Have histologically or cytologically confirmed locally advanced (and not a candidate for definitive therapy) or metastatic NSCLC disease (Stage IIIB or IV) or other solid tumors. For all cohorts except Expansion Cohort 7, the locally advanced or metastatic disease is NSCLC. For Expansion Cohort 7, the locally advanced or metastatic disease is any solid tumor other than NSCLC.
2. Must have sufficient tumor tissue available for analysis.
3. Must have measurable disease by response evaluation criteria in solid tumors (RECIST) v1.1.
4. Male or female adult participants (aged 18 years or older, or as defined per local regulations).
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1.
6. Minimum life expectancy of 3 months or more.
7. Adequate organ function at baseline.
8. Normal QT interval on screening electrocardiogram (ECG), defined as QT interval corrected (Fridericia) (QTcF) of less than or equal to (≤ ) 450 millisecond (ms) in males or ≤ 470 ms in females.
9. Willingness and ability to comply with scheduled visits and study procedures.

Part 1: Dose Escalation Cohort Specific Inclusion Criteria:

1. Refractory to standard available therapies.

Part 2: Expansion Cohort 1 Specific Inclusion Criteria:

1. Have a documented EGFR in-frame exon 20 insertion by a local test.
2. Previously treated with one or more regimens of systemic therapy for locally advanced or metastatic disease.
3. Prior treatment with an EGFR TKI is allowed unless the participants had an objective response and subsequent progression as assessed by the investigator or treating physician.

Expansion Cohort 2 Specific Inclusion Criteria:

1. Have one of the following documented by a local test:

   1. A HER2 exon 20 insertion;
   2. An activating point mutation in HER2.
2. Previously treated with one or more regimens of systemic therapy for locally advanced or metastatic disease.
3. With an EGFR exon 20 insertion: Prior treatment with a pan-HER TKI (example, afatinib, neratinib, or dacomitinib) is allowed unless the participants had an objective response and subsequent progression as assessed by the investigator or treating physician.

Part 2: Expansion Cohort 3 Specific Inclusion Criteria:

1. Have one of the following documented by a local test:

   1. An EGFR exon 20 insertion;
   2. A HER2 exon 20 insertion;
   3. An activating point mutation in HER2.
2. Previously treated with one or more regimen of systemic therapy for locally advanced or metastatic disease.
3. For participants with an EGFR exon 20 insertion: prior treatment with an EGFR TKI is allowed unless the participants had an objective response and subsequent progression as assessed by the investigator or treating physician.
4. For participants with a HER2 exon 20 insertion or HER2 activating point mutation: prior treatment with a pan-HER TKI (example, afatinib, neratinib, or dacomitinib) is allowed unless the participants had an objective response and subsequent progression as assessed by the investigator or treating physician during treatment with that prior TKI.
5. Have either previously untreated intracranial CNS metastases or previously treated intracranial CNS metastases with radiologically documented new or progressing CNS lesions.
6. Have at least one target (that is, measurable) intracranial CNS lesion (greater than or equal to [ ≥ ]10 millimeter [mm] in longest diameter by contrast enhanced magnetic resonance imaging [MRI]).

Part 2: Expansion Cohort 4 Specific Inclusion Criteria:

1. Have one of the following documented by a local test: an activating mutation in EGFR including exon 19 deletions or exon 21 L858R substitution (with or without T790M), or an uncommon activating mutation other than exon 20 insertion including, but not limited to, G719X (where X is any other amino acid), S768I, L861Q, or L861R.
2. Treatment naive for locally advanced or metastatic disease or previously treated with one or more regimens of systemic therapy for locally advanced or metastatic disease.

Part 2: Expansion Cohort 5 Specific Inclusion Criteria:

NSCLC participants with EGFR exon 20 activating insertions, who have previously shown an objective response to an EGFR TKI and subsequently progressed, without active CNS metastases.

1. Have a documented EGFR in-frame exon 20 insertion by a local test.
2. Previously treated with one or more regimens of systemic therapy for locally advanced or metastatic disease.
3. Previously showed an objective response to an EGFR TKI, and subsequently progressed as assessed by the investigator or treating physician.

Part 2: Expansion Cohort 6 Specific Inclusion Criteria:

NSCLC participants with EGFR exon 20 activating insertions, who have not received prior systemic anticancer treatment for locally advanced or metastatic disease, without active CNS metastases.

1. Have a documented EGFR in-frame exon 20 insertion by a local test.
2. No prior systemic treatment for locally advanced or metastatic disease.

Part 2: Expansion Cohort 7 Specific Inclusion Criteria:

Participants with solid tumors other than NSCLC with EGFR/HER2 mutations against which TAK-788 is active, without active CNS metastases.

1. Have a solid tumor that is not NSCLC, including, but not limited to, bladder/urinary tract cancer, breast cancer, gastric/esophageal cancer, biliary tract cancer, and head and neck cancer.
2. Is refractory to standard therapy.
3. Have EGFR or HER2 mutations, documented by a local test.

Part 3: Extension Cohort Specific Inclusion Criteria:

1. Have a documented EGFR in-frame exon 20 insertion by a local test and sufficient tumor tissue available for central analysis.
2. Must have received at least 1 prior line of therapy for locally advanced or metastatic disease and no more than 2 regimens of systemic anticancer chemotherapies for locally advanced or metastatic disease.

   * Prior treatment with an EGFR TKI is allowed unless the participant had an objective response and subsequent progression as assessed by the investigator or treating physician during treatment with that prior TKI.

Exclusion Criteria:

1. Previously received TAK-788.
2. Received small-molecule anticancer therapy (including cytotoxic chemotherapy, and investigational agents, ≤ 14 days prior to first dose of TAK-788 (except for reversible EGFR TKIs [that is, erlotinib or gefitinib], which are allowed in the dose escalation and expansion cohorts up to 7 days prior to the first dose of TAK-788).
3. Received antineoplastic monoclonal antibodies including immunotherapy within 28 days of the first dose of TAK-788.
4. Have been diagnosed with another primary malignancy other than NSCLC except for adequately treated non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or participants with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.

   Note: This exclusion criteria does not apply to Expansion Cohort 7.
5. Received radiotherapy <=14 days prior to the first dose of TAK-788 or has not recovered from radiotherapy-related toxicities. Palliative radiation administered outside the chest and brain, stereotactic radiosurgery (SRS), and stereotactic body radiotherapy are allowed up to 7 days prior to the first dose
6. Received a moderate or strong CYP4503A inhibitor or moderate or strong CYP3A inducer within 10 days prior to first dose of TAK-788.
7. Have undergone major surgery within 28 days prior to first dose of TAK-788. Minor surgical procedures, such as catheter placement or minimally invasive biopsy, are allowed.
8. Part 1 (dose escalation) and Expansion Cohorts 1 to 3 of Part 2 (expansion phase) only:

   Have symptomatic CNS metastases at screening or asymptomatic disease requiring corticosteroids to control symptoms within 7 days prior to the first dose of TAK-788.

   Part 3 (extension cohort) and Expansion Cohorts 4 to 7 of Part 2 (expansion phase) only:

   Have known active brain metastases (have either previously untreated intracranial CNS metastases or previously treated intracranial CNS metastases with radiologically documented new or progressing CNS lesions). Brain metastases are allowed if they have been treated with surgery and/or radiation and have been stable without requiring corticosteroids to control symptoms within 7 days before the first dose of TAK-788, and have no evidence of new or enlarging brain metastases.
9. Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging) or leptomeningeal disease (symptomatic or asymptomatic).
10. Have significant, uncontrolled, or active cardiovascular disease.
11. Have a known history of uncontrolled hypertension. Participants with hypertension should be under treatment on study entry to control blood pressure.
12. Have prolonged QTcF interval, or being treated with medications known to be associated with the development of torsades de pointes.
13. Have an ongoing or active infection, including but not limited to, the requirement for intravenous (IV) antibiotics, or a known history of human immunodeficiency virus, hepatitis B virus (HBV), or hepatitis C virus (HCV). Testing is not required in the absence of history.
14. Currently have or have a history of interstitial lung disease, radiation pneumonitis that required steroid treatment, or drug-related pneumonitis.
15. Female participants who are lactating and breastfeeding or have a positive urine or serum pregnancy test during the screening period.

    Note: Female participants who are lactating will be eligible if they discontinue breastfeeding.
16. Have gastrointestinal illness or disorder that could affect oral absorption of TAK-788.
17. Have any condition or illness that, in the opinion of the investigator, might compromise participant safety or interfere with the evaluation of the safety of the drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2016-06-16 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Part 1, Dose Escalation Component: Recommended Phase 2 Dose (RP2D) of Orally Administered TAK-788 | Cycle 1 (Cycle length is equal to [=] 28 days)
Part 2, Expansion Cohorts 1, 2, 4, 5 and 7: Confirmed Objective Response Rate (ORR) Assessed by the Investigator | Up to 36 months after first dose
Part 2, Expansion Cohort 3: Intracranial ORR (iORR) Assessed by Independent Review Committee (IRC) | Up to 36 months after first dose
Part 2, Expansion Cohort 6: Confirmed ORR Assessed by IRC | Up to 36 months after first dose
Part 3, Extension Cohort: Confirmed ORR Assessed by IRC | Up to 36 months after first dose

SECONDARY OUTCOMES:
Part 1, Dose Escalation Component: Dose Limiting Toxicities (DLTs) of TAK-788 | Cycle 1 (Cycle length=28 days)
Part 1, Dose Escalation Component: Maximum Tolerated Dose (MTD) of TAK-788 | Cycle 1 (Cycle length=28 days)
Parts 1 and 2, Dose Escalation and Expansion Cohorts: Cmax; Maximum Observed Concentration of TAK-788 and its Metabolites | Cycle 1 Day 1 and Cycle 2 Day 1 (cycle length=28 days for Parts 1 and 2)
Parts 1 and 2, Dose Escalation and Expansion Cohorts: Tmax; Time of First Occurrence of Maximum Plasma Concentration (Cmax) of TAK-788 and its Metabolites | Cycle 1 Day 1 and Cycle 2 Day 1 (cycle length=28 days for Parts 1 and 2)
Parts 1 and 2, Dose Escalation and Expansion Cohorts: AUC 24; Area Under the Concentration-time Curve from Time Zero to 24 hours for TAK-788 and its Metabolites | Cycle 1 Day 1 and Cycle 2 Day 1 (cycle length=28 days for Parts 1 and 2)
Parts 1 and 2, Dose Escalation and Expansion Cohorts: AUCt: Area Under the Concentration-time Curve from Time Zero to Time t for TAK-788 and its Metabolites | Cycle 1 Day 1 and Cycle 2 Day 1 (cycle length=28 days for Parts 1 and 2)
Parts 1 and 2, Dose Escalation and Expansion Cohorts: RAC (Cmax): Accumulation Ratio Based on Cmax of TAK-788 and its Metabolites | Cycle 1 Day 1 and Cycle 2 Day 1 (cycle length=28 days for Parts 1 and 2)
Parts 1 and 2, Dose Escalation and Expansion Cohorts: RAC (AUC): Accumulation Ratio Based on AUC of TAK-788 and its Metabolites | Cycle 1 Day 1 and Cycle 2 Day 1 (cycle length=28 days for Parts 1 and 2)
Part 2, Expansion Cohorts 1, 2, 3, 4, 5, and 7: Confirmed ORR as Assessed by IRC | Up to 36 months after first dose
Part 2, Expansion Cohorts: Best Overall Response as Assessed by the Investigator and IRC | Up to 36 months after first dose
Part 2, Expansion Cohorts: Best Target Lesion Response as Assessed by the Investigator and IRC | Up to 36 months after first dose
Parts 2 and 3, Expansion and Extension Cohorts: Duration of Response as Assessed by the Investigator and IRC | Up to 36 months after first dose
Parts 2 and 3, Expansion and Extension Cohorts: Disease Control Rate (DCR) as Assessed by the Investigator and IRC | Up to 36 months after first dose
Part 2 and 3, Expansion and Extension Cohorts: Time to Response as Assessed by the Investigator and IRC | Up to 36 months after first dose
Parts 2 and 3, Expansion and Extension Cohorts: Progression Free Survival (PFS) as Assessed by the Investigator and IRC | Up to 36 months after first dose
Parts 2 and 3, Expansion and Extension Cohorts: Overall Survival (OS) | Up to 36 months after first dose
Part 2, Expansion Cohort 3: Duration of Intracranial Response (iDOR) | up to 36 months after first dose
Part 2, Expansion Cohort 3: Intracranial PFS (iPFS) | up to 36 months after first dose
Part 2, Expansion Cohorts 6: Confirmed ORR as Assessed by the Investigator | Up to 36 months after first dose
Part 3, Extension Cohort: Confirmed ORR as Assessed by the Investigator | Up to 36 months after first dose
Part 3, Number of Participants With Patient-reported Symptoms (Lung Cancer), Functioning, and Health-related Quality of Life (HRQoL) Based on European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-core 30 (EORTC QLQ-C30) | Up to 30 days after last dose of drug (approximately up to 37 months)
Part 3, Extension Cohort: Number of Participants With Patient-reported Symptoms (Lung Cancer), Functioning, and health-related Global Quality of Life (HRQoL) Based on Quality of Life Questionnaire Lung Cancer Module-13 (QLQ-LC13) | Up to 30 days after last dose of drug (approximately up to 37 months)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (62):
- United States (36):
  - Brookwood Medical Center, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - The Oncology Institute of Hope and Innovation - West Tucson, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center - Duarte, Duarte, California
  - Compassionate Cancer Care - Fountain Valley, Fountain Valley, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Pacific Shores Medical Group-Long Beach Elm, Long Beach, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - University of California Irvine Health Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Center - Palo Alto, Palo Alto, California
  - SLO Oncology and Hematology Health Center, San Luis Obispo, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - The University of Chicago Medicine, Chicago, Illinois
  - Investigative Clinical Research - Indiana, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Siteman Cancer Center - Washington University Medical Campus, St Louis, Missouri
  - Atlantic Health - Morristown Medical Center, Morristown, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Thompson Oncology Group - Knoxville - Downtown, Knoxville, Tennessee
  - SCRI - Tennessee Oncology - Nashville - Centennial, Nashville, Tennessee
  - University of Virginia Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Lumi Research, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- China (5):
  - Peking University Cancer Hospital/Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
- Germany (2):
  - Thoraxklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - HELIOS Klinikum Emil von Behring, Berlin
- Italy (2):
  - Istituto Di Ricovero E Cura A Carattere Scientifico - Istituto Europeo Di Oncologia, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
- Japan (4):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kindai University Hospital, Ōsaka-sayama, Osaka
- In Situ Global Clinical Trials Network, Manatí, Puerto Rico
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - Complejo Hospitalario Universitario A Coruna, A Coruña, LA Coruna
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan, Tainan CITY
  - National Taiwan University Hospital - YunLin Branch, Douliu, Yunlin
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- The Royal Marsden NHS Foundation Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Ou SI, Lin HM, Hong JL, Yin Y, Jin S, Lin J, Mehta M, Zhang P, Nguyen D, Neal JW. Comparative effectiveness of mobocertinib and standard of care in patients with NSCLC with EGFR exon 20 insertion mutations: An indirect comparison. Lung Cancer. 2023 May;179:107186. doi: 10.1016/j.lungcan.2023.107186. Epub 2023 Apr 1. PMID 37075617
- [Derived] Christopoulos P, Prawitz T, Hong JL, Lin HM, Hernandez L, Jin S, Tan M, Proskorovsky I, Lin J, Zhang P, Patel JD, Ou SI, Thomas M, Stenzinger A. Indirect comparison of mobocertinib and real-world therapies for pre-treated non-small cell lung cancer with EGFR exon 20 insertion mutations. Lung Cancer. 2023 May;179:107191. doi: 10.1016/j.lungcan.2023.107191. Epub 2023 Apr 8. PMID 37058788
- [Derived] Ou SI, Hong JL, Christopoulos P, Lin HM, Vincent S, Churchill EN, Soeda J, Kazdal D, Stenzinger A, Thomas M. Distribution and Detectability of EGFR Exon 20 Insertion Variants in NSCLC. J Thorac Oncol. 2023 Jun;18(6):744-754. doi: 10.1016/j.jtho.2023.01.086. Epub 2023 Feb 3. PMID 36738930
- [Derived] Yang JC, Zhou C, Janne PA, Ramalingam SS, Kim TM, Riely GJ, Spira AI, Piotrowska Z, Mekhail T, Garcia Campelo MR, Felip E, Bazhenova L, Jin S, Kaur M, Diderichsen PM, Gupta N, Bunn V, Lin J, N Churchill E, Mehta M, Nguyen D. Characterization and management of adverse events observed with mobocertinib (TAK-788) treatment for EGFR exon 20 insertion-positive non-small cell lung cancer. Expert Rev Anticancer Ther. 2023 Jan;23(1):95-106. doi: 10.1080/14737140.2023.2157815. Epub 2022 Dec 28. PMID 36537204
- [Derived] Duke ES, Stapleford L, Drezner N, Amatya AK, Mishra-Kalyani PS, Shen YL, Maxfield K, Zirkelbach JF, Bi Y, Liu J, Zhang X, Wang H, Yang Y, Zheng N, Reece K, Wearne E, Glen JJ, Ojofeitimi I, Scepura B, Nair A, Bikkavilli RK, Ghosh S, Philip R, Pazdur R, Beaver JA, Singh H, Donoghue M. FDA Approval Summary: Mobocertinib for Metastatic Non-Small Cell Lung Cancer with EGFR Exon 20 Insertion Mutations. Clin Cancer Res. 2023 Feb 1;29(3):508-512. doi: 10.1158/1078-0432.CCR-22-2072. PMID 36112541
- [Derived] Zhou C, Ramalingam SS, Kim TM, Kim SW, Yang JC, Riely GJ, Mekhail T, Nguyen D, Garcia Campelo MR, Felip E, Vincent S, Jin S, Griffin C, Bunn V, Lin J, Lin HM, Mehta M, Janne PA. Treatment Outcomes and Safety of Mobocertinib in Platinum-Pretreated Patients With EGFR Exon 20 Insertion-Positive Metastatic Non-Small Cell Lung Cancer: A Phase 1/2 Open-label Nonrandomized Clinical Trial. JAMA Oncol. 2021 Dec 1;7(12):e214761. doi: 10.1001/jamaoncol.2021.4761. Epub 2021 Dec 16. PMID 34647988
- [Derived] Han H, Li S, Chen T, Fitzgerald M, Liu S, Peng C, Tang KH, Cao S, Chouitar J, Wu J, Peng D, Deng J, Gao Z, Baker TE, Li F, Zhang H, Pan Y, Ding H, Hu H, Pyon V, Thakurdin C, Papadopoulos E, Tang S, Gonzalvez F, Chen H, Rivera VM, Brake R, Vincent S, Wong KK. Targeting HER2 Exon 20 Insertion-Mutant Lung Adenocarcinoma with a Novel Tyrosine Kinase Inhibitor Mobocertinib. Cancer Res. 2021 Oct 15;81(20):5311-5324. doi: 10.1158/0008-5472.CAN-21-1526. Epub 2021 Aug 11. PMID 34380634
- [Derived] Riely GJ, Neal JW, Camidge DR, Spira AI, Piotrowska Z, Costa DB, Tsao AS, Patel JD, Gadgeel SM, Bazhenova L, Zhu VW, West HL, Mekhail T, Gentzler RD, Nguyen D, Vincent S, Zhang S, Lin J, Bunn V, Jin S, Li S, Janne PA. Activity and Safety of Mobocertinib (TAK-788) in Previously Treated Non-Small Cell Lung Cancer with EGFR Exon 20 Insertion Mutations from a Phase I/II Trial. Cancer Discov. 2021 Jul;11(7):1688-1699. doi: 10.1158/2159-8290.CD-20-1598. Epub 2021 Feb 25. PMID 33632775
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b601a4db2bf003ab492fd